CLINICAL TRIAL: NCT03105089
Title: Impact of Variable Types of Preconditioning Upon the Inotrope Score in Adult Patients, Undergoing Cardiac Surgery
Brief Title: Effect of Cardiac Preconditioning Upon the Inotrope Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00009910
Record Dates: First submitted 2017-04-02; First posted 2017-04-07 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Open Heart Surgery; Preconditioning
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ischemic preconditioning (Active Comparator): ischemic preconditioning will be done after induction and before cardiopulmonary bypass by inflation the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3cycles
  Interventions: Procedure: ischemic preconditioning
- control (No Intervention): no intervention will be done

INTERVENTIONS:
Procedure: ischemic preconditioning — ) ischemic preconditioning will be done after induction and before cardiopulmonary bypass by inflation the cuff of blood pressure above 200mmhg in the lower limb every 5 min for 3cycles
  Arms: ischemic preconditioning

SUMMARY:
preconditioning of no debate has a valuable effect upon myocardial protection . pre-cardiopulmonary bypass pre-conditioning , suspected to have a role upon postoperative inotropic support

DETAILED DESCRIPTION:
Preconditioning (PC) of the heart occurs when brief exposure to a stimulus protects the heart from subsequent ischemia. PC stimulus may be ( ischemic ;pharmacologic or Physical) Pharmacological pc may be induced by variable agents e.g. (Sevoflurane ;isoflorane, opioids etc ) Ischemic pc includes local ;remote and the idea is temporary interruption of blood supply to the organ so that liberation of protective mediators occurs The liberated mediators have favorable effects not only upon the myocardium But ;it extend to protect other organs against inflammatory activation ;ischemia reperfusion injury Inotropic score IS is already an evident predictor of postoperative cardiac mobidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* valve replacement surgery
* ASA grade 2 or 3

Exclusion Criteria:

* emergency surgery
* - poor general conditions
* impaired hepatic or renal function
* peripheral vascular disease
* patient refusal

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
inotropic score | 48 hours

SECONDARY OUTCOMES:
renal function | 2 dyas
  serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided